CLINICAL TRIAL: NCT04440865
Title: Impact of Artificial Intelligence Genius® System-assisted Colonoscopy vs. Standard Colonoscopy on Adenoma Detection Rate in Routine Practice: a Prospective Randomized Controlled Trial
Brief Title: Impact of Artificial Intelligence Genius® System-assisted Colonoscopy vs. Standard Colonoscopy (COLO-GENIUS)
Acronym: COLO-GENIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Paris-Bercy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COLO-GENIUS
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Colonic Polyp; Colonoscopy; Artificial Intelligence; Colonic Adenoma; Colonic Neoplasms
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Arm 1- Standard colonoscopy Arm 2- Colonoscopy assisted by Genius® system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Standard colonoscopy (Active Comparator): Standard colonoscopy is performed
  Interventions: Other: Standard Colonoscopy
- Arm 2- Colonoscopy assisted by Genius (Active Comparator): Colonoscopy assisted by Genius artificial intelligence system is performed
  Interventions: Other: Genius® System-assisted Colonoscopy

INTERVENTIONS:
Other: Genius® System-assisted Colonoscopy — Genius® Intelligence System is used to assist Colonoscopy
  Arms: Arm 2- Colonoscopy assisted by Genius
Other: Standard Colonoscopy — Standard Colonoscopy without Genius® Intelligence System is performed
  Arms: Arm 1- Standard colonoscopy

SUMMARY:
This controlled-randomized trial compares the artificial intelligence Genius® system assisted (Genius+) to standard (Genius-) colonoscopy.

The aim of this study was to evaluate the impact of Genius® system on ADR in routine colonoscopy. The secondary aims will be the impact of Genius® system on polyp detection rate (PDR), serrated polyp detection rate (SPDR), advanced neoplasia detection rate (ANDR), mean number of polyps (MNP), polyp type and localization, and operator type (according to basal ADR).

DETAILED DESCRIPTION:
Any patient seen by gastroenterologists working in the endoscopy unit and meeting the inclusion criteria may be recruited.

The patient will be offered to participate in the study. The information form as well as the consent, will be given to the patient for a good understanding of the study and the investigator in charge of the patient gives all the additional explanations necessary for this good understanding (but of the study, the course, risks and benefits).

A period of reflection will be left to the patient or his family to make a free decision whether or not to participate in the study.

After the consent to participate will be signed by the gastroenterologist and the patient, the patient will be randomized. The use of the Genius® system will depend on the randomization that will be performed at the start of the colonoscopy.

This randomization will be done in the computer examination room using the randomization software.

The patient will therefore be randomized into 2 groups:

Arm 1- Standard colonoscopy Arm 2- Colonoscopy assisted by Genius® system

A comparison of the two groups standard colonoscopy vs colonoscopy assisted by Genius® system will be made as following:

A-Main criterion:

- Adenoma detection rate (ADR)

B-Secondary criteria:

Polyps detection rate (PDR) Proximal serrated polyps detection rate (PSPDR) Neoplasia detection rate (NDR) Mean number of polyps (MNP) Mean number of adenomas (MNA) Factors associated with ADR

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for total colonoscopic exploration, during the period study
* Patient over or equal to 18 years
* ASA 1, ASA 2, ASA 3
* No participation in another clinical study
* Certificate of non opposition signed

Exclusion Criteria:

* Patient under 18 years old
* ASA 4, ASA 5
* Pregnant woman
* Patient with coagulation abnormalities preventing polypectomy: prothrombin level <50%, Platelets <50000 / mm3, effective anti-coagulation in progress, clopidogrel in progress.
* Patient referred for resection of a known polyp
* Inflammatory bowel disease
* Known colonic stenosis
* Diverticulitis less than 6 weeks old
* Patient unable to give consent or protected by law
* Opposition expressed for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | 1 day
  percentage of colonoscopy with one or more adenoma of the colon

SECONDARY OUTCOMES:
Advanced Neoplasia Detection Rate (ANDR) | 1 day
  percentage of colonoscopy with one or more advanced neoplasia of the colon
Proximal Serrated Polyp Detection Rate (PSPDR) | 1 day
  percentage of colonoscopy with one or more serrated polyp of the colon
Polyp Detection Rate (PDR) | 1 day
  percentage of colonoscopy with one or more polyp of the colon
The factors influencing the Adenoma Detection Rate (ADR) | 1 day
  Withdrawal time (in seconds): time of exploration from the caecum to the anal verge
The factors influencing the Adenoma Detection Rate (ADR) | 1 day
  Boston scale (0 to 9)
Time to reach caecum (sec) | 1 day
  Time to reach caecum from the beginning of the procedure (in seconds)
Caecal intubation rate (%) | 1 day
  Caecal intubation rate (complete colonoscopy)
Morbidity: perforation rate (%) | 7 days after procedure
  Perforation rates (%)
Morbidity: bleeding rate (%) | 7 days after procedure
  Bleeding rates (%)

CONTACTS AND LOCATIONS:
Overall Officials: David Karsenti, MD, Study Director — Clinique Paris-Bercy
Locations (1):
- Clinique Paris-Bercy, Charenton-le-Pont, France

REFERENCES:
- [Derived] Karsenti D, Tharsis G, Perrot B, Cattan P, Percie du Sert A, Venezia F, Zrihen E, Gillet A, Lab JP, Tordjman G, Cavicchi M. Effect of real-time computer-aided detection of colorectal adenoma in routine colonoscopy (COLO-GENIUS): a single-centre randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Aug;8(8):726-734. doi: 10.1016/S2468-1253(23)00104-8. Epub 2023 Jun 1. PMID 37269872